CLINICAL TRIAL: NCT03254056
Title: The Effects of Fascial Closure Techniques on Post-Operative Pain in Gynecologic Laparoscopic Surgery
Brief Title: Fascial Closure Techniques Post-Operative Pain Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Hasan Onur Topçu, Associate Professor, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZTB1
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Post-operative Pain; Fascial Closure
Keywords: fascial closure device; laparoscopic surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Technique (Active Comparator): The edges of the fascia will be hold by the surgical instruments. The fascial defect will be repaired by using devices which are generated for laparotomy operations.
  Interventions: Procedure: Conventional technique
- Berci Technique (Active Comparator): This instrument facilitates full thickness abdominal wall closure under the view of laparoscopic optic.
  Interventions: Procedure: Berci technique

INTERVENTIONS:
Procedure: Conventional technique — Conventional technique: In this group; S-retractors will be used to visualize the fascia and a single interrupted stitch will be placed using 0-vicryl suture.
  Arms: Conventional Technique
Procedure: Berci technique — Berci group: In this group; the fascial incision will be closed with the fascial closure device, (Berci Fascial Closure instrument) using 1 interrupted stitch with 0-vicryl suture.
  Arms: Berci Technique

SUMMARY:
This study compares post-operative incisional pain on post-operative days 1 and 7 who will undergo gynecologic laparoscopic operations. Half of participants will undergo conventional fascial closure, while the other will undergo fascial closure by Berci Fascial Closure (Karl Storz, Belgium).

DETAILED DESCRIPTION:
Studies have demonstrated that laparoscopic surgery has numerous advantages over laparotomy. The patients who undergo laparoscopic surgery acquired fewer doses of analgesics than who undergo laparotomy. This point is also one of the advantages of the laparoscopic surgery. The fascia closure in fascial defects larger than 10 mm diameters in laparoscopic surgery is an important issue. Incisional hernias may occur after laparoscopic surgery. The surgeons prefer the techniques in fascial closure which is more safe and cause less pain. In current study, investigators aim to compare the post-operative incisional pain in two different techniques in gynecologic laparoscopic surgery; conventional versus by 'Berci Fascial Closure'.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Ability to understand the inform consent
3. No conversion from laparoscopy to laparotomy

Exclusion Criteria:

1. No-ability to understand the inform consent
2. Conversion to laparotomy from laparoscopy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Post-operative incisional pain | 24 hours after fascial closure closure
  Visual Analog Scale
Post-operative incisional pain | 7 days after fascial closure closure
  Visual Analog Scale

SECONDARY OUTCOMES:
Time for fascial closure | Intraoperative
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yaprak Üstün, Prof, Study Chair — University of Health Sciences, Zekai Tahir Burak Women's Health Health Research and Practice Center
Locations (1):
- Zekai Tahir Burak Women Health Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lyapis A, Ulrich A, LaMonica R, Kuo CL, Kaye L, Luciano D. Does the Difference in Fascial Closure Technique Affect Postoperative Pain? J Minim Invasive Gynecol. 2017 Nov-Dec;24(7):1190-1194. doi: 10.1016/j.jmig.2017.07.020. Epub 2017 Jul 27. PMID 28757438
- [Result] Williams CP, Rosen MJ, Jin J, McGee MF, Schomisch SJ, Ponsky J. Objective analysis of the accuracy and efficacy of a novel fascial closure device. Surg Innov. 2008 Dec;15(4):307-11. doi: 10.1177/1553350608327168. PMID 19036733
- [Result] Elashry OM, Nakada SY, Wolf JS Jr, Figenshau RS, McDougall EM, Clayman RV. Comparative clinical study of port-closure techniques following laparoscopic surgery. J Am Coll Surg. 1996 Oct;183(4):335-44. PMID 8843262